CLINICAL TRIAL: NCT04121104
Title: Electrodermal Activity and Respiration in Patients Treated With Spinal Cord Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, Principal Investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SWEAT
Record Dates: First submitted 2019-05-04; First posted 2019-10-09 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Spinal cord stimulation; Electrodermal activity
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCS off (Experimental)
  Interventions: Other: SCS is switched off
- SCS on (Experimental)
  Interventions: Other: SCS is switched on

INTERVENTIONS:
Other: SCS is switched off — Spinal cord stimulator is switched off for 12 hours
  Arms: SCS off
Other: SCS is switched on — Spinal cord stimulator is on
  Arms: SCS on

SUMMARY:
This study is investigating skin conductance and respiration during on and off states of the spinal cord stimulator, in patients with failed back surgery syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old.
* Diagnosis of FBSS (Failed conservative treatments for pain including but not limited to pharmacological therapy and physical therapy) and currently being treated with spinal cord stimulation.
* Cognitive and language functioning enabling coherent communication between the examiner and the participant.

Exclusion Criteria:

* Patients with impaired skin integrity at the fingers.
* Patients with major psychiatric problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Skin conductance changes | Two times on the same day; once while SCS is switched off and once while SCS is switched on. Total study duration lasts one day.]
  The investigators will examine the difference in skin conductance between both measurements (SCS on versus SCS off)
Respiration rate | Two times on the same day; once while SCS is switched off and once while SCS is switched on. Total study duration lasts one day.]
  The investigators will examine the difference in respiration rate between both measurements (SCS on versus SCS off)

SECONDARY OUTCOMES:
Pain intensity scores using the Visual Analogue Scale | Two times on the same day; once while SCS is switched off and once while SCS is switched on. Total study duration lasts one day.]
  Pain intensity score on that time on a Visual Analogue Scale (VAS) ranging from zero (no pain) towards 10 (worst possible pain) for the pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Moens, Prof. dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - Clinique Ste Elisabeth, Verviers